CLINICAL TRIAL: NCT00062491
Title: Phase 2 Trial of Karenitecin (BNP1350) in Patients With Malignant Melanoma
Brief Title: Study of Karenitecin (BNP1350) to Treat Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioNumerik Pharmaceuticals, Inc. (Industry)
Collaborators: Crown Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTN23106
Record Dates: First submitted 2003-06-06; First posted 2003-06-12 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Melanoma; Neoplasm
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — cositecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Karenitecin (BNP1350)
  Interventions: Drug: Karenitecin (BNP1350)

INTERVENTIONS:
Drug: Karenitecin (BNP1350) — Karenitecn (1.0 mg/m2) administered as a single daily 60-minute intravenous infusion for 5 consecutive days repeated every 21 days (1 treatment cycle). Patients who respond (CR< PR, SD) can continue treatment for 6 cycles, unless unacceptable toxicity develops. Treatment will be discontinued if progressive disease or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Karenitecin (BNP1350) as a treatment for Malignant Melanoma.

ELIGIBILITY:
* Confirmed diagnosis of malignant melanoma
* Measurable disease
* Granulocytes ≥1,500/µl, Platelets ≥100,000/µl, Creatinine ≤ULN, Bilirubin ≤1.5 mg/dl, AST ≤2.5 x ULN
* No prior treatment with other camptothecin drug.
* ≥ 21 days since completion of prior chemotherapy, ≥6 weeks since prior Mitomycin-C
* ECOG Performance Status 0-1
* Negative pregnancy test for female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2002-05; Primary Completion 2003-06 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Overall Response | start of treatment until progressive disease

SECONDARY OUTCOMES:
Objective Tumor Response Rate | Start of treatment to date of response
Duration of Response | Date of response to date of progressive disease
Overall Survival | Randomization to date of death from any cause
Progression Free Survival | Randomization to disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- For Information call 210-614-1701 for a site near you, Tampa, Florida, United States